CLINICAL TRIAL: NCT02701582
Title: Goal-Directed Intraoperative Fluid Management Using FloTrac© Monitoring in High-Risk Neurosurgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-01043
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Intracranial Aneurysm; Brain Edema; Scoliosis; Surgery
MeSH Terms: conditions — Intracranial Aneurysm; Brain Edema; Scoliosis | interventions — Phenylephrine; Pseudoephedrine; Acetaminophen; Epinephrine; Albumins; HES 130-0.4; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Goal Directed Therapy (Experimental): Flotrack monitor is connected and based on what anesthesiologist sees and following study algorithm, anesthesiologist chooses: Phenylephrine, Epinephrine , volume resuscitation (fluids, including normal saline, albumin, voluven and packed red blood cells) and no intervention.
  Interventions: Drug: Phenylephrine; Drug: Epinephrine; Other: Albumin; Other: Voluven; Other: Normal Saline; Other: Packed Red Blood Cells; Device: FloTrac Monitor
- Control Group (Active Comparator): FloTrac monitor is connected, but he anesthesiologist will not be able to see the monitor although the data will be collected and stored for analysis. Anesthesiologist will be given a study algorithm to follow for the duration of the surgery, and based on it will choose: Phenylephrine, Epinephrine , volume resuscitation (fluids, including normal saline, albumin, voluven and packed red blood cells) and no intervention.
  Interventions: Drug: Phenylephrine; Drug: Epinephrine; Other: Albumin; Other: Voluven; Other: Normal Saline; Other: Packed Red Blood Cells; Device: FloTrac Monitor

INTERVENTIONS:
Drug: Phenylephrine — if Mean arterial pressure (MAP) is < = 65, Stroke volume variation (SVV) < 13 and Cardiac Index is >=2.2 Phenylephrine is administered
  Other Names: Sudafed; Neo-Synephrine; SudoGest
Drug: Epinephrine — if Mean arterial pressure (MAP) is < = 65, Stroke volume variation (SVV) < 13 and Cardiac Index is < 2.2 Epinephrine is administered
  Other Names: EpiPen; Adrenaclick; Medihaler-Epi
Other: Albumin — if Mean arterial pressure (MAP) is < = 65, Stroke volume variation (SVV) > = 13, fluids are administered --OR-- if Mean arterial pressure (MAP) is > 65, Stroke volume variation (SVV) > = 13 and Cardiac Index is <2.2 fluids are administered.
Other: Voluven — if Mean arterial pressure (MAP) is < = 65, Stroke volume variation (SVV) > = 13, fluids are administered --OR-- if Mean arterial pressure (MAP) is > 65, Stroke volume variation (SVV) > = 13 and Cardiac Index is <2.2 fluids are administered.
Other: Normal Saline — if Mean arterial pressure (MAP) is < = 65, Stroke volume variation (SVV) > = 13, fluids are administered --OR-- if Mean arterial pressure (MAP) is > 65, Stroke volume variation (SVV) > = 13 and Cardiac Index is <2.2 fluids are administered.
Other: Packed Red Blood Cells — if Mean arterial pressure (MAP) is < = 65, Stroke volume variation (SVV) > = 13, fluids are administered --OR-- if Mean arterial pressure (MAP) is > 65, Stroke volume variation (SVV) > = 13 and Cardiac Index is <2.2 fluids are administered.
Device: FloTrac Monitor — FloTrac monitor is connected for all patients, but only visible to the anesthesiologist for half. Based on a decision tree and the data from monitor, choices of interventions are used.

SUMMARY:
This is a prospective, randomized controlled trial to determine if using FloTrac/EV1000 system in neurosurgical patients undergoing craniotomies for aneurysm repair or tumor resection complicated by cerebral edema, or complex spinal surgery including multi-level scoliosis correction, is a more effective way of monitoring fluid.

DETAILED DESCRIPTION:
We hypothesize that the ability to assess volume status and fluid responsiveness with information gained from Edwards FloTrac/EV1000 system coupled with a goal-directed therapy fluid management algorithm can make a difference in patient outcomes. Our specific aims are:

* Demonstrate goal-directed therapy (GDT) in fluid management improves peri-operative fluid balance
* Demonstrate GDT improves pulmonary function and organ oxygenation
* Demonstrate GDT reduces necessary therapeutic interventions in the peri- operative period
* Demonstrate GDT reduces hypotensive episodes in the peri-operative period

Outcomes

We will study the consequences of goal-directed fluid therapy that employs use of dynamic indicators seen on FloTrac/EV1000 system by measuring the following:

* Pulmonary status

  * Time to extubation
  * Alveolar-arterial (A-a) gradient of oxygen
  * Requirements for supplemental oxygen
* Organ oxygenation

  * Serum lactate
  * Arterial blood gas values (pH, HCO3, CO2, O2)
* Length of stay (LOS)

  * In hospital, defined as time from operation start to eligibility for discharge from hospital according to surgeon in accordance with pre-define criteria
  * In ICU/PACU, defined as time from operation end to eligibility for discharge from intensive care according to attending intensivist in accordance with pre- define criteria
* Fluid Balance

  * Inputs and outputs (I/Os) of all measurable fluids (i.e. blood, crystalloid, colloid) in peri-operative period, through and including duration of intensive care or the next 24-48 hours after completion of surgery
  * Drugs administered for fluid management (i.e. mannitol, vasopressors)
  * Pre-operative and post-operative body weights and twice-daily weights via bed weights
* Hypotension

  * Number, duration and severity (i.e. minimum blood pressure) of hypotensive episode, defined as MAP <65

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical patients with concerns for decreased intracranial compliance;
* Orthopedic spine patients;
* Patients scheduled to undergo neurosurgical interventions that include any of the following will be eligible: intracranial aneurysm repair; or, major spine surgery.

Exclusion Criteria:

* Patients with permanent cardiac arrhythmias;
* Patients with severe aortic regurgitation;
* Patients with intra-aortic balloon pump (IABP);
* Patients undergoing emergency surgery; and,
* Women who are pregnant and/or nursing will be excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bloom, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were prescreened and slate was given to PI for approval. Patients were approached in pre-op on day of surgery in a private setting. Study was discussed with them and questions were answered. If interested, they signed consent.
  Study team began screening patients after receiving IRB approval. The first patient was consented on 3/13/14.
Groups:
- Goal Directed Therapy: Anesthesiologists have access to monitor, so they can follow the study algorithm, for the duration of the surgery. Anesthesiologist may choose to discontinue the study algorithm at any time based on his or her best clinical judgment. Clinical judgment can and must always override the study protocol if discrepancy exists. If this occurs, the patient would be considered to fail the protocol, and be considered in a separate group in data analysis.
  FloTrac Sensor: Care based on algorithm and device.
- Control Group: FloTrac will be connected to the monitor but anesthesiologists will not be able to see the monitor. The data will be collected and stored for analysis. Anesthesiologist will choose from the same drug and fluid options used in the FloTrac (GDT) group (phenylephrine, epinephrine, normal saline, albumin, Voluven), but to be used in accordance with their best clinical judgment without the aid of the FloTrac data. If a discrepancy exists, the attending anesthesiologist may choose to use other therapies not included in the GDT protocol, in accordance with their best clinical judgment. If this happens, the subject would be considered to fail the protocol, and be considered in a separate group in data analysis.
  FloTrac Algorithm Not Visible: Standard of Care
Period: Overall Study
Arm/Group | Goal Directed Therapy | Control Group
Started | 35 | 33
Completed | 33 | 33
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Goal DIrected Therapy: Anesthesiologist will be able to see the dynamic indicators, and will be given a study algorithm to follow, based on the trending data, for the duration of the surgery. Anesthesiologist may choose to discontinue the study algorithm at any time based on his or her best clinical judgment. Clinical judgment can and must always override the study protocol if discrepancy exists. If this occurs, the patient would be considered to fail the protocol, and be considered in a separate group in data analysis.
  FloTrac Sensor: Care based on algorithm and device.
- Control Group: FloTrac will be connected to the monitor, the anesthesiologist will not be able to see the monitor although the data will be collected and stored for analysis. Anesthesiologist will be asked to choose from the same drug and fluid options used in the GDT group (phenylephrine, epinephrine, normal saline, albumin, Voluven), but to be used in accordance with their best clinical judgment without the aid of FloTrac data. If a discrepancy exists, the attending anesthesiologist may choose to use other therapies not included in the GDT protocol, in accordance with their best clinical judgment. If this happens, the subject would be considered to fail the protocol, and be considered in a separate group in data analysis.
  FloTrac Algorithm Not Visible: Standard of Care
- Total: Total of all reporting groups
Arm/Group | Goal DIrected Therapy | Control Group | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 12 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 22 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 26 | 24 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of ICU Stays Greater Than 1.5 Days
Description: the sum of ICU stays greater than the 1.5 Days eligibility for discharge from hospital according to the surgeon, over the course of 20 Days
Time Frame: 20 Days
Measure: Number (95% Confidence Interval); unit: Number of ICU Stays greater that 1.5 Day
Groups:
- Goal Directed Therapy: FloTrac monitor visible, care based on algorithm and device.
- Control Group: FloTrac monitor not visible, standard of care
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
Number of ICU Stays greater that 1.5 Day | 13 [7 to 19] | 20 [14 to 26]

2. Secondary Outcome: Creatinine Change
Description: Change in creatinine in the 72 hour post-op period (mg/dL)
Time Frame: Baseline and 72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
mg/dL | -0.04 (0.25) | -0.13 (0.16)

3. Other Pre Specified Outcome: Pulmonary Status as Measured by the Number of Participants Who Require Supplemental Oxygen
Description: We looked at the number of patients who required supplemental oxygen within the first 24 hours after surgery.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
Participants | 17 | 25

4. Other Pre Specified Outcome: Organ Oxygenation as Measured by Serum Lactate
Description: Serum lactate levels, as measured in mmol/L, in patients during the first 24 hours after surgery.
Time Frame: Baseline and 24 Hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
mmol/L | 2.0 (1.15) | 1.75 (1.04)

5. Other Pre Specified Outcome: Organ Oxygenation as Measured by Arterial Blood Gas Values
Description: Patient's organ oxygenation as measured by base deficit mEq/L, during the first 24 hours after surgery.
Time Frame: Baseline and 1 day
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
mEq/L | 3.55 (3.96) | 4.75 (4.45)

6. Other Pre Specified Outcome: Fluid Balance Measured by Inputs and Outputs (I/Os) of All Measurable Fluid in Peri-operative Period
Description: Fluid balance measured by I/Os of all fluid in the peri-op period during the first 12 hours after the subject's surgery.
Time Frame: Baseline and 12 Hours
Population: Data not collected. This outcome measure was not included by PI in reported results
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
ml/kg | NA (NA) — This outcome measure was not included by PI in reported results. This outcome measure was not analyzed and is not being provided by PI. | NA (NA) — This outcome measure was not included by PI in reported results. This outcome measure was not analyzed and is not being provided by PI.

7. Other Pre Specified Outcome: Patients Requiring Fluid Bolus for Management
Description: Number of patients who received fluid boluses in the first 24 hours post-op
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
Participants | 7 | 6

8. Other Pre Specified Outcome: Number of Patients Treated for Hypotension With Phenylephrine Drip
Description: The number of patients on a phenylephrine drip within 24 hours post-op.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 4

9. Other Pre Specified Outcome: Area Under Curve of MAP Below 65
Description: Hypotension as measured by area under the curve of MAP less than 65.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: mmHG x minutes
Arm/Group | Goal Directed Therapy | Control Group
Number analyzed (Participants) | 33 | 33
mmHG x minutes | -65.06 (63.89) | -61.88 (64.23)

ADVERSE EVENTS:
Groups:
- FloTrac Sensor: FloTrac monitor visible, care based on algorithm and device.
Arm/Group | FloTrac Sensor | Control Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No